CLINICAL TRIAL: NCT02743650
Title: Pilot Study of Sodium Bicarbonate in Generally Healthy People With Low Bicarbonate
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties identifying subjects who were qualified to participate in the study
Sponsor: University of Utah (Other)
Collaborators: The University of Utah Center on Aging (Unknown)
Responsible Party: Principal Investigator, Kalani Raphael, Principal Investigator, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 81006
Record Dates: First submitted 2016-04-06; First posted 2016-04-19 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Chronic Kidney Disease
Keywords: Low Serum Bicarbonate Level; Sodium Bicarbonate
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sodium Bicarbonate (Experimental): All participants will receive oral sodium bicarbonate for 6 weeks (On-treatment period). After the 6 week visit, participants will stop taking sodium bicarbonate and return for a final visit 4 weeks later (Off-treatment period).
  The initial dose of sodium bicarbonate prescribed is 0.3 mEq/kg/d. If a subject meets the protocol criteria, the dose will be increased to 0.6 mEq/kg/d. Half the dose will be taken by mouth in the morning and the other half in the evening.
  Interventions: Dietary Supplement: Sodium bicarbonate

INTERVENTIONS:
Dietary Supplement: Sodium bicarbonate — The initial dose of sodium bicarbonate is 0.3 mEq/kg/d. If a subject meets the protocol criteria, the dose will be increased to 0.6 mEq/kg/d.

SUMMARY:
The goal of this pilot study is to determine whether oral sodium bicarbonate can raise low serum bicarbonate concentration in people without chronic kidney disease (CKD). Participants will take sodium bicarbonate for six weeks, followed by a four week washout period.

DETAILED DESCRIPTION:
CKD affects 25 million Americans and the risks of cardiovascular morbidity, hospitalizations, and death are substantially higher for people with CKD. Furthermore, 6% of the total Medicare budget is spent on 600,000 people with end-stage renal disease. Thus, CKD is highly prevalent, associates with poor outcomes, and is a tremendous financial burden to society.

Apart from treating hypertension and diabetes, there are no therapies that prevent CKD. However, results from two studies have found that low serum bicarbonate levels increase risk of developing CKD, which suggests that normalizing low serum bicarbonate may prevent CKD.

One way to raise low serum bicarbonate is by taking sodium bicarbonate. Whether sodium bicarbonate, which is commonly prescribed to raise low serum bicarbonate in people with CKD, can raise low bicarbonate in people without CKD is uncertain because the reason bicarbonate is low in people without CKD is unclear. This is because low bicarbonate by itself cannot distinguish whether the acid-base abnormality is primary metabolic acidosis or respiratory alkalosis. The former process is readily corrected with alkali. However, the administration of alkali in the latter situation may not raise bicarbonate concentration.

Therefore, the purpose of this pilot study is to determine whether oral sodium bicarbonate can raise low serum bicarbonate in people without renal disease.

The study is a single-arm open label study of 15 individuals without CKD with low serum bicarbonate concentration. The study duration is 10 weeks. After completing the baseline visit, participants will take oral sodium bicarbonate (initial dose level: 0.3 milliequivalents per kilogram per day (mEq/kg/d) for 6 weeks (On-treatment period), followed by a 4 week Off-treatment period. Serum concentrations of sodium bicarbonate will be tested during the treatment period, at the end of the On-treatment period (Week 6) and at the end of the Off-treatment period (Week 10).

ELIGIBILITY:
Inclusion Criteria:

* Estimated glomerular filtration rate (eGFR) ≥ 60 ml/min/1.73m2
* Urinary albumin/creatinine ratio < 30 mg/gm
* Serum bicarbonate ≤ 23 mEq/L (average of the two most recent measurements within the past year)
* Age ≥ 50 years

Exclusion Criteria:

* Blood pressure ≥ 160/100 mm Hg
* Serum potassium < 3.5 mEq/L
* New York Heart Association Class 3 or 4 heart failure symptoms
* Chronic oxygen therapy
* Chronic obstructive pulmonary disease requiring daily bronchodilator or prednisone therapy
* Weight ≥ 160 kg
* Use of sodium bicarbonate, sodium citrate, potassium citrate, or potassium bicarbonate within the previous two weeks.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-02; Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Change in serum bicarbonate concentration from baseline to 6 weeks | Baseline and 6 weeks
  Comparison of pre-intervention serum bicarbonate levels to week 6 levels following treatment with oral sodium bicarbonate.

SECONDARY OUTCOMES:
Change in serum bicarbonate concentration after 4 weeks of stopping sodium bicarbonate treatment | Baseline, 6 weeks and 10 weeks
  Comparison of serum bicarbonate levels four weeks after discontinuing oral sodium bicarbonate treatment to pre-intervention (baseline) and immediate post-treatment (week 6) serum bicarbonate levels.

CONTACTS AND LOCATIONS:
Overall Officials: Kalani L Raphael, MD, Principal Investigator — VA Salt Lake City Healthcare System
Locations (1):
- VA Salt Lake City Healthcare System, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldenstein L, Driver TH, Fried LF, Rifkin DE, Patel KV, Yenchek RH, Harris TB, Kritchevsky SB, Newman AB, Sarnak MJ, Shlipak MG, Ix JH; Health ABC Study Investigators. Serum bicarbonate concentrations and kidney disease progression in community-living elders: the Health, Aging, and Body Composition (Health ABC) Study. Am J Kidney Dis. 2014 Oct;64(4):542-9. doi: 10.1053/j.ajkd.2014.05.009. Epub 2014 Jun 18. PMID 24953890
- [Background] Driver TH, Shlipak MG, Katz R, Goldenstein L, Sarnak MJ, Hoofnagle AN, Siscovick DS, Kestenbaum B, de Boer IH, Ix JH. Low serum bicarbonate and kidney function decline: the Multi-Ethnic Study of Atherosclerosis (MESA). Am J Kidney Dis. 2014 Oct;64(4):534-41. doi: 10.1053/j.ajkd.2014.05.008. Epub 2014 Jun 18. PMID 24953891